CLINICAL TRIAL: NCT04325217
Title: Post-marketing Surveillance on Long Term Use of Ofev Capsules in Systemic Scleroderma Associated Interstitial Lung Disease (SSc-ILD) in Japan
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0387
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients newly initiating Ofev®/Nintedanib Capsules
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Capsules
  Other Names: Ofev®

SUMMARY:
The primary objective is to confirm the incidence of adverse drug reactions (focus on gastrointestinal symptoms including diarrhoea and nausea) to Ofev Capsules seen in clinical trials with real world data generated in patients with SSc-ILD.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Japan with SSc-ILD who are prescribed with Ofev Capsules and have never been treated with Ofev Capsules before enrolment will be included.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: As this is a non-interventional study, no specific treatment is mandated or withheld from the patients. No limitations are set up on background factors and their concomitant drugs in use of actual medical practice.
Sampling Method: Probability Sample
Enrollment: 586 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) | up to 3 years and 9 months
  Focus on gastrointestinal symptoms including diarrhea and nausea

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com